CLINICAL TRIAL: NCT05716698
Title: Health Evaluation of Mushrooms withVitamin D2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N202111054
Record Dates: First submitted 2023-01-09; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-02

CONDITIONS: Healthy
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): no Pleurotus citrinopileatus intervention
- D2 10ug Pleurotus citrinopileatus Group (Experimental): took D2 10ug Pleurotus citrinopileatus per day for a total of 4 weeks.
  Interventions: Dietary Supplement: Pleurotus citrinopileatus after bio-optics (10 ug group)
- D2 100ug Pleurotus citrinopileatus Group (Experimental): took D2 100ug Pleurotus citrinopileatus per day for a total of 4 weeks.
  Interventions: Dietary Supplement: Pleurotus citrinopileatus after bio-optics (100 ug group)

INTERVENTIONS:
Dietary Supplement: Pleurotus citrinopileatus after bio-optics (10 ug group) — The participants took D2 10ug per day for a total of 4 weeks.
  Arms: D2 10ug Pleurotus citrinopileatus Group
Dietary Supplement: Pleurotus citrinopileatus after bio-optics (100 ug group) — The participants took D2 100ug per day for a total of 4 weeks.
  Arms: D2 100ug Pleurotus citrinopileatus Group

SUMMARY:
Although Taiwan has plenty of sunshine, the intake of vitamin D and the concentration of 25(OH)D in the blood are low. Ingestion of mushrooms and extracts rich in D2 can increase the nutritional source of vitamin D. The purpose of this study is to evaluate the intake of D2 mushrooms and extracts in humans to achieve the effective concentration of 25(OH)D in the serum and recommendations for health improvement.

DETAILED DESCRIPTION:
The subjects were divided into 3 groups: no mushroom intervention, intervention with D2 10ug Pleurotus citrinopileatus after bio-optics optimization (low dose group) or intervention with D2 100ug Pleurotus citrinopileatus after bio-optics optimization (high dose group). The low-dose group took D2 10ug per day, and the high-dose group received D2 100ug per day for a total of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy human

Exclusion Criteria:

1. Any acute disease, such as infection, stroke, myocardial infarction or major surgery within three months, upper or lower gastrointestinal bleeding, blood pressure, and poor blood sugar control will be excluded.
2. Chronic diseases, such as malignant tumors, infection with human immunodeficiency virus (HIV) and related diseases, liver cirrhosis, or those with liver function exceeding 3 times the normal value (more than 120 IU/L), renal function (Cr) more than 2.5 mg /dl, chronic anemia (Hb <9 g/dl), metabolic diseases except diabetes (such as thyroid/parathyroid dysfunction), and those who have undergone abdominal surgery to cause intestinal sticking are excluded.
3. Women who are pregnant or breastfeeding will be excluded.
4. Those who use steroids, supplements with vitamin D-containing dietary supplements and hormones will be excluded.
5. Those with blood 25(OH)D concentration > 30 ng/ml will be excluded.
6. Those who are unwilling to fill out the consent form and refuse the questionnaire survey.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 25OHD at week 4 | Baseline and week 4
  The participants' blood was taken to analyze the concentration of 25OHD to compare the changes between baseline and 4 weeks later. 25OHD concentration standard is:
  25OHD < 20 ng/ml: deficiency 20 ng/ml < 25OHD < 30 ng/ml: Insufficiency 25OHD > 30 ng/ml: Normal

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Han Lin, MS, Principal Investigator — Office of Human Research, Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No